CLINICAL TRIAL: NCT06104280
Title: Medications for Opioid Use Disorder Differentially Modulate Intrinsically Photosensitive Retinal Ganglion Cell Function, Sleep, and Circadian Rhythms: Implications for Treatment (MOUD)
Brief Title: Medications for Opioid Use Disorder Photosensitive Retinal Ganglion Cell Function, Sleep, and Circadian Rhythms: Implications for Treatment
Acronym: MOUD
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Karen Cropsey, Professor, University of Alabama at Birmingham
Other Study IDs: IRB-300011499; R01DA059471-01 (NIH)
Record Dates: First submitted 2023-09-19; First posted 2023-10-27 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Opioid Use Disorder; Sleep Disturbance
Keywords: opioid use disorder; sleep; circadian rhythms; sleep disruption
MeSH Terms: conditions — Opioid-Related Disorders; Parasomnias | interventions — Ecological Momentary Assessment; Actigraphy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- MOUD therapy methadone: 50 methadone participants
  Interventions: Other: Post-Illumination Pupillary Response (PIPR); Other: Polysomnography; Other: Multiple Sleep Latency Test; Behavioral: Ecological Momentary Assessments; Device: Actigraphy; Other: DLMO; Other: Melatonin Suppression Test
- MOUD therapy buprenorphine: 50 buprenorphine participants
  Interventions: Other: Post-Illumination Pupillary Response (PIPR); Other: Polysomnography; Other: Multiple Sleep Latency Test; Behavioral: Ecological Momentary Assessments; Device: Actigraphy; Other: DLMO; Other: Melatonin Suppression Test
- MOUD therapy extended-release naltrexone: 50 extended-release naltrexone (XR-NTX) participants
  Interventions: Other: Post-Illumination Pupillary Response (PIPR); Other: Polysomnography; Other: Multiple Sleep Latency Test; Behavioral: Ecological Momentary Assessments; Device: Actigraphy; Other: DLMO; Other: Melatonin Suppression Test
- Non-opioid using controls: non-opioid using controls
  Interventions: Other: Post-Illumination Pupillary Response (PIPR); Other: Polysomnography; Other: Multiple Sleep Latency Test; Behavioral: Ecological Momentary Assessments; Device: Actigraphy; Other: DLMO; Other: Melatonin Suppression Test

INTERVENTIONS:
Other: Post-Illumination Pupillary Response (PIPR) — The PIPR is measured in six, 80-s test periods in which the stimulus, either Blue (470 nm) or Red (623 nm), is presented to the dilated eye while the pupil response of the un-dilated eye is measured (consensual pupil response
  Other Names: PIPR
Other: Polysomnography — Measure electroencephalography (EEG), electrooculography (EOG), electromyography (EMG), electrocardiography (ECG), respiratory channels (effort and nasal pressure), and oxygen saturation.
  Other Names: PSG
Other: Multiple Sleep Latency Test — Assist in the diagnosis of disorders of hypersomnolence,63 it is also used in research to quantify daytime sleepiness and serves as a more objective measure of daytime sleepiness than self-report questionnaires
  Other Names: MSLT
Behavioral: Ecological Momentary Assessments — Morning after overnight Visit 2, participants will complete ecological momentary assessments (EMAs) over a 10-day assessment period. Using EMA through the InsightTM mHealth platform to capture momentary craving, withdrawal and mood states across 10 days among persons who smoke and nonsmokers prior to an overnight procedures. Participants will complete morning and evening sleep diaries via the EMA InsightTM mHealth platform self-reported sleep and wake information, fatigue, naps, opioid craving and withdrawal.
  Other Names: EMA
Device: Actigraphy — 7-day actigraphy period will be used to determine the habitual sleep start and wake times. The CamNTech MotionWatch8 (Cambridge, UK) is a solid-state piezo-electric accelerometer that collects data on activity (i.e., arm motion) and ambient light.Actigraphy data are downloaded from the MotionWatch8 into the software (MotionWare) for analysis, management, and exportation. Bed and wake times will be entered by the subjects via a REDCap link and this information coupled with the sleep diary reports will be entered to determine sleep intervals. Algorithms in the Motion Watch 8 software will determine sleep start, sleep end, total sleep time (duration), sleep quality, sleep efficiency, wake after sleep onset, and sleep fragmentation
Other: DLMO — Participants will be given an evening meal and then be accompanied to the UAB Highlands Hospital Sleep Unit by 5:30pm. The sleep unit allows for strict control of light exposure (< 5 lux at eye level), room temperature and oral intake factors that could alter melatonin levels.Participants will be allowed to sleep in darkness until 8:00am, at which time they will be provided transportation.We will also bank frozen samples taken prior to the light exposure for later calculation of the Dim Light Melatonin Onset (DLMO), a circadian phase estimate.
  Other Names: Dim Light Melatonin Onset
Other: Melatonin Suppression Test — The sleep unit allows for strict control of light exposure (< 5 lux at eye level), room temperature and oral intake factors that could alter melatonin levels. Participants will be asked to refrain from caffeine consumption 12 hours before reporting to the sleep unit and will provide 2-3 ml of saliva every 30 minutes starting at 6:00pm and ending after the light exposure. For melatonin suppression, 2-hours light exposure will begin 2 hours before the calculated mid-sleep time. Collection saliva samples 1-h, 30-min, and immediately before the light exposure and every 30 min throughout exposure. Samples will be centrifuged and frozen/stored at -20ºC until assay and remaining samples stored at -80ºC. Melatonin levels will be assayed via the Buhlmann Direct Saliva Melatonin. Melatonin suppression will be calculated as the percent decrease from the sample taken immediately prior to the light exposure

SUMMARY:
Opioid use disorder (OUD) is a treatable medical illness with three medications FDA approved for treatment. However, persons with OUD report significant sleep disturbance, even when treated with medications for opioid use disorder, leading to high rates of relapse. In this project, we will investigate a special set of photosensitive neurons in the retina as an underlying mechanism for circadian rhythm and sleep disturbance from opioid use and medications for OUD that could lead to novel intervention and improve treatment outcomes.

DETAILED DESCRIPTION:
Three medications for OUD (MOUD) are FDA-approved and regularly used to treat OUD: methadone, buprenorphine, and extended-release naltrexone (XR-NTX). However, persons who use opioids, including those prescribed MOUDs, report sleep disruption. In addition to the sleep centers of the brain, mu opioid receptors (MORs) are also expressed in the retina (including the human retina), specifically in ganglion cells that are critically important for non-image forming photoreception including circadian regulation of sleep-wake behavior. Pre-clinical studies show that activation of MORs on these intrinsically photosensitive retinal ganglion cells (ipRGCs) reduces the electrophysiological response to light, impacting critical ipRGC functions such as synchronization of sleep-wake behavior and circadian rhythms to light (photoentrainment), light-induced melatonin suppression, and the post-illumination pupillary reflex (PIPR). Together, these results suggest that activation of MORs in the ipRGCs by opioid use and/or MOUDs may impair downstream ipRGC functions. This multi-disciplinary study will examine the novel overarching hypothesis that persistent alterations in sleep/wake behavior in OUD patients undergoing treatment are mediated by impaired ipRGC function, and biomarkers of this pathway can predict recovery and relapse. Three aims will be tested in a sample of 200 participants, 150 of whom will be engaged in MOUD therapy (e.g., 50 each on methadone, buprenorphine, and XR-NTX, respectively) and 50 of whom will be non-opioid using control participants. Aim 1 will test the hypothesis that MOUD differentially impacts function of ipRGC responses. Aim 2 will examine whether MOUD differentially impacts daytime sleepiness, daily sleep-wake behavior, sleep architecture, and sleep-disordered breathing. Finally, Aim 3 will determine if ipRGC function predicts opioid relapse among MOUD groups at 1-, 3- and 6- month follow-up. Compared to non-opioid using controls or persons receiving an opioid antagonist (XR-NTX), we predict that participants who are receiving an agonist (methadone) or partial-agonist (buprenorphine) MOUD will have the most ipRGC interference, as evidenced by reduced PIPR, attenuated light-induced melatonin suppression, reduced circadian rhythmic amplitude, increased sleep latency, and increased sleep fragmentation. Importantly, we hypothesize that impaired ipRGC function will predict worse treatment outcomes as indicated by opioid use by 6-month follow-up. Finally, an exploratory aim will examine whether the MOUD groups show different relationships between opioid craving/withdrawal symptoms and sleep-wake behavior over a 10-day assessment of the participants' daily lives within the normal environment. The results of this study will be highly significant because it would support the use of the pupillary response to light and other indicators of ipRGC function as novel biomarkers to predict the response and outcomes to MOUDs.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18+)
2. prescribed one of three medications for opioid use disorder (methadone, XR-NTX, buprenorphine) or healthy control
3. stable on MOUD (no dose change) for the past month
4. positive on urine drug screen (UDS) for buprenorphine or methadone if prescribed those medications

Exclusion Criteria:

1. eye disease reported by history or noted on exam including disease of the anterior and posterior segment of the eye, cataracts, retinopathy, glaucoma, cataracts, amblyopia, scotoma, color or night blindness, corneal pathologies, macular degeneration, or retinitis pigmentosa;
2. acutely suicidal, manic, intoxicated, or otherwise not stable enough to provide informed consent
3. self-reported use of illicit opioids, stimulants (prescribed or illicit), or benzodiazepines/sedative/hypnotics in the past month
4. alcohol or cannabis use disorder measured as severe on The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) Checklist
5. positive on UDS for illicit opioids (e.g., morphine, oxycodone, fentanyl),stimulants, benzodiazepines/sedative/hypnotics
6. shift workers who work outside normal 7 a.m. to 6 p.m. hours, according to the National Institute of Occupational Safety and Health (NIOSH)
7. persons diagnosed with narcolepsy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study involves people who are receiving one of three medications for opioid use disorder (methadone, buprenorphine or naltrexone) or healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2028-12-28 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Aim 1: Post-Illumination Pupillary Response (PIPR) | 45 minutes
  10-day at home actigraphy and ecological momentary assessments (EMA period), participants will be scheduled for Visit 3. Upon arrival, the non-dominant eye is dilated with Tropicamide 0.5% and Phenylephrine 2.5% (this lower-than-normal dilation dosage will be effective for the duration of the experiment but will fully dissipate within ~6 hours). Subjects are then seated in a dimly lit room (< 5 lux, background light) for 30 minute to dark adapt and to ensure complete pupil dilation prior to the study. The PIPR is measured in six, 80-second test periods in which the stimulus, either Blue (470 nm) or Red (623 nm), is presented to the dilated eye while the pupil response of the un-dilated eye is measured (consensual pupil response). During a test period, after an initial 20-second fixation period, the stimulus is presented for 1 second followed by a 60-second fixation period. The red stimulus primarily serves as a control for any nonspecific influences on the PIPR.
Aim 2: Polysomnography | 2 night PSG
  Polysomnography (PSG)110: To avoid potential first-night effects often observed with PSG, participants will undergo two consecutive nights of PSG, scheduled to begin according to their habitual sleep/wake times. PSG will be conducted in dedicated research rooms located at the University of Alabama at Birmingham Sleep/Wake Disorders Center at Highlands Hospital (refer to Sleep and Circadian Research Core LOS). Trained staff will attach electrodes to measure electroencephalography (EEG), electrooculography (EOG), electromyography (EMG), electrocardiography (ECG), respiratory channels (effort and nasal pressure), and oxygen saturation. The values of the EEG, EOG, EMG, ECG respiratory channels, and oxygen saturation will be combined to report a single PSG value.
Aim 3: Number of Participants Multiple Sleep Latency Test | 2 night PSG
  On the morning following the second night of PSG, participants will undergo an MSLT following standardized guidelines. Briefly, the multiple sleep latency test (MSLT) consists of 5 nap opportunities that occur every two hours with the first nap beginning 1.5 to 3 hours after the end of the PSG (in this case, after the end of the 2nd night of PSG).
Aim 4: Number of Participants with Relapse | 6-month follow up
  Self reported drug cravings, and self-reported withdrawal symptoms by 6-month follow up.Self-reported and urine drug screen confirmed drug use.

SECONDARY OUTCOMES:
Dim Light Melatonin Onset (DLMO) | 12 hours
  Samples taken prior to the light exposure for later calculation of the Dim Light Melatonin Onset (DLMO)
Melatonin suppression test | 12 hours
  Melatonin suppression test, actigraphy parameters (rhythmic amplitude, inter-daily stability, intra-daily variation, sleep fragmentation, sleep efficiency, sleep duration, mid-sleep time, and wake after sleep onset), and sleep architecture (PSG). provide 2-3 ml of saliva every 30 min starting at 6:00pm and ending after the light exposure.Participants will be seated in a chair in front of a white light source lights will be calibrated for intensity and spectral distribution at eye level with a PR-670 spectrophotometer). During the light exposure, participants will be allowed to watch an unexciting movie on a 15-inch iPad tablet. Collect saliva samples 1-h, 30-min, and immediately before the light exposure and every 30 min throughout exposure. After the last sample, participants will be allowed to sleep in darkness until 8:00 am

CONTACTS AND LOCATIONS:
Overall Officials: Karen Cropsey, PsyD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No